CLINICAL TRIAL: NCT05589909
Title: Performance of Interleukin-27 Cord Blood Level as A Biomarker Predicating Early Onset Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Wael Seliem, Professor of Pediatrics and Neonatology, Mansoura University Children Hospital
Other Study IDs: R.22.03.1667
Record Dates: First submitted 2022-06-12; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Neonatal Sepsis, Early-Onset
Keywords: Early onset neonatal sepsis, Procalcitonin, Interleukin-27.
MeSH Terms: conditions — Neonatal Sepsis | interventions — Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection Group: Both suspected and confirmed sepsis occurred ≤72 hours after delivery were counted as cases of EONS.
  Interventions: Diagnostic Test: IL27, PCT, CRP, Blood culture
- None Infection Group: No evidence clinical or laboratory of infection
  Interventions: Diagnostic Test: IL27, PCT, CRP, Blood culture

INTERVENTIONS:
Diagnostic Test: IL27, PCT, CRP, Blood culture — magnetic bead multiplex platform

SUMMARY:
Neonatal sepsis still considered as one of the major causes of mortality and morbidity during the neonatal period due to high vulnerability of that age group. The blood culture is considered as the gold standard for diagnosis of bacterial sepsis, however in early onset neonatal sepsis (EONS) the inability to isolate a microbial pathogen does not exclude sepsis. The reason behind the high number of culture-negative cases is not clear and might be attributed to low levels of bacteremia or small volumes of blood obtained from sick infants. Also maternal antibiotic treatment before or during delivery may theoretically mask detection of bacteremia in the newborn. In addition these cultures have a 48-72 hours delay to obtain results. Therefore, the combination of clinical assessment and laboratory biomarkers currently are the bases for diagnosis of neonatal sepsis.

Recently interleukin-27 (IL-27) has been looked at as another candidate biomarker in the serum for diagnosis of sepsis in both adult and children. Interleukin-27 (IL-27), a novel member of the IL-12 family, was first discovered in 2002. IL- 27 is primarily synthesized by antigen-presenting cells, and it is widely expressed in a myriad of cells, including placental trophoblast cells. Although multiple studies have reported IL-27 as an essential regulator of immune response and inflammation, its precise role in the immune response is still disputable.

Conventionally, IL-27 has been envisaged as a potent promoter of inflammation. When first discovered, it was characterized as a promoting factor in the rapid initiation of inflammatory responses, processing the ability to stimulate the rapid expansion of naïve CD4+T and then the production of IFN-?, which has been demonstrated by various subsequent studies.

The aim of this study was to evaluate the usage of elevated IL-27 in cord blood as an early predictor biomarker for EONS.

DETAILED DESCRIPTION:
A prospective study will be conducted in the neonatal intensive care unit (NICU), Mansoura University Children Hospital -over a period of one year. The study subjects will include all newborn infants born to pregnant women with one or more of antenatal risk factors for sepsis including maternal fever, prolonged rupture of membranes with leakage of amniotic fluid preceding the onset of labor for 18 hours or more, presence of chorioamnionitis or evidence of maternal colonization with group B streptococcus (GBS). Prematurity was defined as gestational age of 36+6 weeks and less.

Blood samples for biomarkers detection will be collected from the umbilical artery after clamping the umbilical cords before delivery of the placenta. The blood will be collected in ethylene diamine tetra-acetic acid-containing tubes from each infant for immunological detection of IL-27, procalcitonin and C-reactive protein.

For neonatal blood culture, blood samples will be collected from each neonate, before starting any antimicrobial treatment, by venous puncture from a peripheral vein for blood culture. About 1 mL of blood will be directly inoculated into a pediatric blood culture bottle and sent to the Medical Microbiology and Immunology Department, Mansoura University, Egypt for subsequent microbiological processing. Obtained bacterial isolates will be identified by standard microbiological techniques

ELIGIBILITY:
Inclusion Criteria:

* All newborn infants born to pregnant women who had one or more of antenatal risk factors for sepsis. on or evidence of maternal colonization with group B streptococcus (GBS).

Exclusion Criteria: None

-

Ages: 0 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: These risk factors included maternal fever, prolonged rupture of membranes with leaking amniotic fluid 18 hours or more before delivery, maternal bacterial infection including urinary tract infection or evidence of maternal colonization with group B streptococcus (GBS).
Sampling Method: Non-Probability Sample
Enrollment: 548 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-22 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of IL27, PCT and CRP levels in umbilical cord blood | 6 months
  comparison between 2 groups

SECONDARY OUTCOMES:
Measurement of IL27, PCT and CRP levels in blood after 24 hours | 6 months
  comparison between 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
If not used in extended research work